CLINICAL TRIAL: NCT05050708
Title: Risikofaktorer for Postoperativ Smerte og Kvalme Etter Dagkirurgisk Gynekologisk Laparoskopi
Brief Title: Riskfactors of Post-operative Pain and Nausea After Ambulatory Gynaecological Laparocopy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, professor, Oslo University Hospital
Other Study IDs: Gyn.smerte.op.risiko.21
Record Dates: First submitted 2021-08-23; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Postoperative Nausea
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient interview — Patient will be interviewed pre-operatively and at 24 hrs post-opartively

SUMMARY:
Patient due for elective, ambulatory gynaecological laparoscopy will be screened peri-operatively for known and potential risk factors of postoperative pain and nausea/vomiting.

The actual incidence and severity of pain and nausea/vomiting will be recorded during th 0-24 hr intervall after end of surgery, as well as the doses of all drugs, given for either prophylaxis or treatment

ELIGIBILITY:
Inclusion Criteria:

* Elective adult patients due for planned ambulatory gynaecological laparoscopy
* Must be able to speak and write in Norwegian language

Exclusion Criteria:

* Patients who, for some reason, is transferred to non-ambulatory (same day discharge) care.
* Patients who, for some reason, have a change in surgical procedure from laparoscopy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self representation of gender identity
Study Population: Adult females
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 0-24 hours
  Numerical Ratings Score (NRS) Scale 0-10, 10 is worst
postoperative nausea | 0-24 hours
  yes/no, Numerical Rating Score (NRS), Scale 0-10, 10 is worst

SECONDARY OUTCOMES:
Peri-operative nausea risk score | preop, 0-24 hours post-operatively
  Apfel score, 0-4 (4 is maximal risk).Based on a number of registrations, such as: smoking status, postoperative opioid effects, smoking status, travel sickness, previous nause or vomiting after surgery/anaesthesia
Peri-operative pain risk score | preop, 0-24 hours
  Based on a number of registrations, such as: age, sosio-economic status, pre-op pain, pre-op use of opioids, pre-op anxiety or depression, pre-op catastrophizing, pre-op expectations, type of surgery, type of anaesthesia, lenght/ivasive ness of surgery, peri-op drug consumtion
Post-op fatigue | 0-24 hrs
  Christensen score, 0-10, 10 is maximal fatigue
Post-op function | 0-24hr
  Everyday function
Post-op analgesia consumption | 0-24hr
  number of opioid equivalents consumed
Post-op anti-emetic drug consumption | 0-24hr
  type and dose of ante-emetic medication

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided